CLINICAL TRIAL: NCT03888053
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of Topical BB-101 (rhNEGF) for the Treatment of Diabetic Lower Leg and Foot Ulcers
Brief Title: BB-101 for Treatment of Diabetic Lower Leg and Foot Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blue Blood Biotech Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BB-101-001A
Record Dates: First submitted 2019-02-20; First posted 2019-03-25 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BB-101 Treatment Arm (Active Comparator): BB-101 liquid formulation concentration of 2 µg/mL or 20 µg/mL will be applied on the target lower leg or foot ulcer once a day for 4 consecutive weeks.
  Interventions: Biological: BB-101
- Placebo Arm (Placebo Comparator): Placebo will be applied on the target lower leg or foot ulcer once a day for 4 consecutive weeks.
  Interventions: Biological: BB-101

INTERVENTIONS:
Biological: BB-101 — Within each cohort, 8 subjects will be randomized to receive BB-101 and 4 subjects to receive placebo.

SUMMARY:
This is a randomized, double-blind, placebo-controlled, sequential dose escalation study in diabetic subjects with a diabetic lower leg or foot ulcer. All subjects will receive standard-of-care ulcer treatment from screening through the last study visit.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, sequential dose escalation study in diabetic subjects with a diabetic lower leg or foot ulcer. All subjects will receive standard-of-care ulcer treatment from screening through the last study visit.

The study will be conducted at multiple investigational sites located in Taiwan. Additional sites and countries may be added during the course of the study if required.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 20 years of age and older.
* Type 1 or type 2 diabetes mellitus.
* Glycosylated hemoglobin (HbA1c) of ≤12%.
* A target ulcer on the lower leg or foot that meets the following criteria at screening:

  1. located below knees,
  2. Area of 0.5 - 10.0 cm^2 following sharp debridement , as measured at Visit 1 and confirmed at Visit 2,
  3. Extending through the epidermis and dermis but not involving bone, tendon or ligament,
  4. Present for ≥4 weeks prior to Visit 1 despite appropriate care, and
  5. Ulcer without clinical signs and symptoms of infection.
* Adequate arterial blood supply to the lower leg or foot under study, to be measured either by doppler ultrasonography, ankle brachial pressure index (ABPI) ≥0.70, or toe pressure >30 mmHg.
* Female subjects of childbearing potential must have a negative serum pregnancy test prior to first dose of study medication and must agree to use an effective method of contraception throughout the study. Females who are surgically sterile or have been postmenopausal for at least 1 year (12 consecutive months without menses) are exempted from these criteria. Effective methods of contraception include oral contraceptives, injectable or implantable hormonal methods, intrauterine devices, tubal ligation (if performed more than 1 year prior to screening), or double barrier contraception (e.g., diaphragm+condom).
* Subject agrees to comply with ulcer care regimen for the duration of the study.
* Subject is able to understand and sign an informed consent form and willing to comply with all study procedures.

Exclusion Criteria:

* Clinical signs and symptoms of infection of target ulcer assessed by clinical evaluation (the presence of infection is defined by ≥2 classic findings of inflammation or purulence).
* Presence of cellulitis or gangrene on the lower leg or foot under study.
* Presence of another open ulcer <2 cm away from target ulcer, on the same lower leg or foot.
* Target ulcer on the heel.
* Target ulcer caused primarily by untreated arterial insufficiency or with an etiology not related to diabetes.
* Subjects with ulcers related to an incompletely healed amputation wound.
* Acute or chronic osteomyelitis affecting the area of the target ulcer.
* Any structural deformity of the lower leg or foot under study that would prevent off- loading of the target ulcer, including acute Charcot osteoarthropathy.
* Previous use of a platelet-derived product (e.g., becaplermin) or other growth factors on the target ulcer within 4 weeks prior to Visit 1.
* Previous use of autologous graft or allogeneic graft, or dermal substitute or living skin equivalent (e.g., Dermagraft® or Apligraf®) on the target ulcer or hyperbaric oxygen therapy within 2 weeks prior to Visit 1.
* Use of any topical antimicrobials or enzymatic debridement treatment, to treat the target ulcer within 7 days prior to Visit 1.
* Treatment with systemic corticosteroids other than for inhalation, immunosuppressive agents, radiation therapy, or chemotherapeutic agent within 30 days prior to Visit 1 or likelihood to receive any of these therapies during study participation.
* History of cancer or current cancer, with the exception of adequately treated or excised non-melanoma skin cancer.
* Vasculitis, connective tissue diseases, or any medical conditions known to impair ulcer healing, other than diabetes.
* Sickle cell disease.
* Clinically significant electrocardiogram (ECG) abnormality, as determined by the Investigator.
* Any of the following laboratory results at screening: serum creatinine >2.5 mg/dL; aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2x upper limit of normal (ULN).
* Poor nutritional status (serum albumin < 2.5 g/dL).
* A history of drug or alcohol abuse that could compromise compliance or safety.
* History of human immunodeficiency virus (HIV) infection.
* Known sensitivity to any component of BB-101 or placebo.
* Participation in a clinical trial of an investigational drug or device within 30 days of study entry.
* Pregnancy, lactation, or plans to become pregnant within 6 months.
* Any social or medical condition that, in the opinion of the Investigator, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
* History of non-compliance with treatment or clinical visit attendance.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of local reactions | 6 weeks
  To assess the incidence of local reactions for target ulcer and surrounding area and record the severity
Incidence and severity of adverse events | 6 weeks
  To assess the incidence of adverse events and record the severity
Incidence of clinical laboratory abnormalities | 6 weeks
  To assess the incidence of clinical laboratory abnormalities
Change from baseline in ECG | 6 weeks
  To assess the change of baseline in ECG
Change from baseline in blood pressure | 6 weeks
  To assess the change of baseline in in blood pressure
Change from baseline in heart rate | 6 weeks
  To assess the change of baseline in heart rate
Change from baseline in body temperature | 6 weeks
  To assess the change of baseline in body temperature
Presence of anti-BB-101 antibodies | 6 weeks
  To assess the immunogenecity for BB-101

SECONDARY OUTCOMES:
Proportion of subjects with target ulcer that heals within the 4-week treatment period | 4 weeks
  complete healing defined as re-epithelialization without drainage and dressing requirement
To evaluate plasma concentration of BB-101 | 4 weeks
  To evaluate plasma concentration of BB-101

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Chen Pan, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan